CLINICAL TRIAL: NCT02229513
Title: Uterine Cooling During Cesarean Delivery to Reduce Blood Loss and Incidence of Postpartum Hemorrhage: A Randomized Controlled Trial
Brief Title: Uterine Cooling During Cesarean Delivery to Reduce Blood Loss and Incidence of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 013-035
Record Dates: First submitted 2014-08-07; First posted 2014-09-01 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2015-12

CONDITIONS: Postpartum Hemorrhage; Uterine Atony
Keywords: postpartum hemorrhage; uterine atony; cesarean section; cesarean hysterectomy; acute blood loss anemia; uterotonics; obstetric hemorrhage; severe hemorrhage; blood transfusion; obstetric emergencies; obstetrics; massive hemorrhage; hemorrhage; uterine cooling
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Normal cesarean technique.
- Uterine Cooling (Experimental): Immediately following delivery of the fetus the uterus will be externalized in the usual fashion and the body of the uterus cephalad to the hysterotomy incision will be wrapped in sterile surgical towels saturated in sterile, iced normal saline. These towels will come from a sterile cooling pot set to 30 degrees Fahrenheit. Iced saline-soaked towels will be kept in place for a minimum of 5 minutes and replaced at the discretion of the attending obstetrician until the hysterotomy is closed and the uterus is replaced into the patient's abdomen.
  Interventions: Procedure: Uterine Cooling

INTERVENTIONS:
Procedure: Uterine Cooling — Immediately following delivery of the fetus the uterus will be externalized in the usual fashion and the body of the uterus cephalad to the hysterotomy incision will be wrapped in sterile surgical towels saturated in sterile, iced normal saline. These towels will come from a sterile cooling pot set to 30 degrees Fahrenheit. Iced saline-soaked towels will be kept in place for a minimum of 5 minutes and replaced at the discretion of the attending obstetrician until the hysterotomy is closed and the uterus is replaced into the patient's abdomen.
  Other Names: Hush Slush Machine
  Arms: Uterine Cooling

SUMMARY:
The objective of the study is to demonstrate whether cooling the uterine smooth muscle during cesarean section (following delivery of the fetus) will promote better uterine contraction and involution resulting in lower blood loss, use of fewer uterotonic medications, and fewer hysterectomies following cesarean section. The investigators suspect that it may.

DETAILED DESCRIPTION:
Study Design:

Patients will be randomly assigned to either the study group or the control group. Patients may receive regional (epidural or spinal/epidural) or general anesthesia.Initially, the investigators plan to enroll 200 subjects, 100 to the study group and 100 to the control group.

Following delivery of the fetus, patients in the study group also will have Pitocin® administered to them according to the usual protocol.Immediately following delivery of the fetus the uterus will be externalized in the usual fashion and the body of the uterus cephalad to the hysterotomy incision will be wrapped in sterile surgical towels saturated in sterile, iced normal saline. These towels will come from a sterile cooling pot set to 30 degrees Fahrenheit. The skin of the abdomen will be draped to prevent contact with the cold towels. Additional uterotonic medications may be given at the discretion of the attending obstetrician.

Iced saline-soaked towels will be kept in place for a minimum of 5 minutes and replaced at the discretion of the attending obstetrician until the hysterotomy is closed and the uterus is replaced into the patient's abdomen. The surface temperature of the uterus will be measured using an infrared thermometer prior to replacing the uterus into the abdomen.

Two surgical suction canisters will be available. Immediately after delivery of the fetus and prior to delivery of the placenta, the amniotic fluid and blood on the surgical field will be aspirated into the first canister. The second suction canister will be used to aspirate blood and fluid until the conclusion of the operation.

At the conclusion of the surgery blood loss will be calculated by measuring the content of blood in the second canister minus the amount of irrigation fluid used, and by weighing the surgical sponges. Average blood loss during cesarean sections has previously been reported as 500 to 1000 cc.

The duration of cooling the uterus will be recorded.

Use and amount of uterotonic medications also will be recorded.

During the surgery the patient's vital signs will be monitored in the usual fashion. Particular attention will be paid to a change in her temperature. Warmed blankets and forced air warming blankets will be used to maintain normothermia, if required.

At the conclusion of the study the amount of blood loss between the control and study groups, and the amount of uterotonic drugs will be calculated and compared. The number of patients in each group who require additional surgeries, e.g. hysterectomy or D&C, will be monitored. Pre-op and post-op hemograms will be compared if obtained at the discretion of the attending obstetrician. Blood product administration will be recorded.

Determination of an ideal temperature of cooling towels is not an objective of the study. We're asking a qualitative question, not a quantitative question at this time.

Study Rationale: The uterus is a smooth muscle whose contraction is modulated most directly by intrinsic or extrinsic oxytocin. During pregnancy the spiral arteries within the uterus and beneath the placenta enlarge to provide adequate perfusion to the placenta. After separation of the placenta the uterine smooth muscle cells contract in a pincer-like action to pinch the spiral arteries closed. When uterine contraction is inadequate (approximately 4-6% of normal pregnancies) the spiral arteries continue to bleed. If not addressed the bleeding can be excessive, even leading to maternal death. Approximately 5-8 out of 1,000 cesarean sections require hysterectomy to control bleeding.

Release of calcium ions from sarcoplasmic reticulum stores is the immediate initiator of contraction, and calcium's diffusion from the muscle filaments and re-uptake by the sarcoplasmic reticulum results in relaxation of contraction. In some smooth muscles cold enhances contraction; perhaps by slowing the re-uptake of calcium. When the usual pharmacologic agents fail to induce adequate contraction of the uterine smooth muscle, the investigators suspect that application of cold may.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant adult women of any gravidity, and gestational duration who present for cesarean section at Baylor University Medical Center in Dallas and who have given informed consent to be in the study.

Exclusion Criteria:

* Women who refuse to be in the study, and women who are unable to consent due to emergent nature of the cesarean section will be excluded. Women who are unable to understand the nature of the study due to mental illness, mental retardation, medical condition, or other communication barrier will be excluded.
* Inability to exteriorize the uterus during c-section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice L Mitchell, MD, Principal Investigator — Baylor University Medical Center Resident
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Uterine Cooling
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Uterine Cooling: Immediately following delivery of the fetus the uterus will be externalized in the usual fashion and the body of the uterus will be wrapped in sterile surgical towels saturated in sterile, iced normal saline. These towels will come from a sterile cooling pot set to 30 degrees Fahrenheit. Iced saline-soaked towels will be kept in place for a minimum of 5 minutes and replaced at the discretion of the attending obstetrician until the hysterotomy is closed and the uterus is replaced into the patient's abdomen.
- Total: Total of all reporting groups
Arm/Group | Control | Uterine Cooling | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (4.8) | 31.7 (5.1) | 30.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 82 | 78 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height (ft) [Mean (Standard Deviation); unit: feet] | 5.4 (0.2) | 5.4 (0.3) | 5.4 (0.3)
Weight (lbs) [Mean (Standard Deviation); unit: pounds] | 200 (49) | 187 (39) | 194 (45)
Gravidity [Mean (Full Range); unit: pregnancies] | 2.5 [1 to 7] | 2.4 [1 to 9] | 2.5 [1 to 9]
Parity [Mean (Full Range); unit: births] | 1.0 [0 to 5] | 1.0 [0 to 4] | 1.0 [0 to 5]
Gestational Age (wks) [Mean (Standard Deviation); unit: weeks] | 38.5 (2.2) | 38.0 (4.2) | 38.3 (3.4)
Fetal Presentation [Number; unit: participants]
  Cephalic | 84 | 83 | 167
  Breech | 14 | 14 | 28
  Transverse | 1 | 2 | 3
  Oblique | 1 | 0 | 1
  Compound | 0 | 1 | 1
Multiple Gestations [Number; unit: participants]
  yes | 11 | 7 | 18
  no | 89 | 93 | 182
Fetal Weight (g) [Mean (Standard Deviation); unit: grams] | 3504 (852) | 3471 (822) | 3488 (835)
Previous Cesareans [Mean (Full Range); unit: cesareans] | 0.8 [0 to 3] | 0.7 [0 to 3] | 0.8 [0 to 3]
Trial of Labor [Number; unit: participants]
  yes | 7 | 16 | 23
  no | 93 | 84 | 177
Pre-op Epidural [Number; unit: participants]
  yes | 9 | 17 | 26
  no | 91 | 83 | 174

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: At the conclusion of the surgery, blood loss will be calculated by measuring the content of blood in the suction canister, and by weighing the surgical sponges. The amount of blood loss in the PACU will be measured by weighing pads.
Time Frame: During surgery and in the PACU (approximately 3 total hours)
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
cc
  Intraoperative blood loss | 616 (411) | 418 (317)
  PACU blood loss | 141 (199) | 106 (170)
  Total blood loss | 756 (462) | 536 (429)

2. Secondary Outcome: Change in Pre- vs Post-operative Hematocrit
Time Frame: 48 hours post operative period
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
percent | 4.3 (3.6) | 4.8 (3.1)

3. Secondary Outcome: Use of Uterotonic Medications
Time Frame: During surgery and in the PACU (approximately 3 total hours)
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 5 | 4
  no | 95 | 96

4. Secondary Outcome: Use of Extra Oxytocin
Time Frame: Intraoperatively
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 1 | 1
  no | 99 | 99

5. Other Pre Specified Outcome: Patient Temperature
Time Frame: Pre-op, Intra-op, Post-Op
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
degrees Fahrenheit
  Pre-operative | 98.3 (0.4) | 98.4 (0.7)
  Intra-operative | 97.7 (1.0) | 97.9 (0.7)
  Post-operative | 97.8 (0.4) | 97.9 (1.0)

6. Other Pre Specified Outcome: Total Time Uterus Wrapped
Time Frame: During hysterotomy repair
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
minutes | 9.3 (4.3) | 9.4 (4.0)

7. Other Pre Specified Outcome: Uterine Temperature After Wrap Removed
Time Frame: Immediately following hysterotomy repair
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
degrees Fahrenheit | 88.3 (3.0) | 75.5 (7.8)

8. Secondary Outcome: Use of Methergine
Time Frame: Intraoperatively
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 2 | 2
  no | 98 | 98

9. Secondary Outcome: Use of Hemabate
Time Frame: Intraoperatively
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 1 | 2
  no | 99 | 98

10. Secondary Outcome: Use of Cytotec
Time Frame: Intraoperatively
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 4 | 3
  no | 96 | 97

11. Secondary Outcome: Bakri Bulb Placement
Time Frame: Intraoperatively
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 3 | 0
  no | 97 | 100

12. Secondary Outcome: Use of Additional Measures to Control Blood Loss, Including Pharmacological and Surgical Interventions
Time Frame: Intraoperatively
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 6 | 5
  no | 94 | 95

13. Secondary Outcome: Requirement of Blood Products
Time Frame: During surgery and in the PACU (approximately 3 total hours)
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 2 | 3
  no | 98 | 97

14. Secondary Outcome: Total Blood Loss Greater Than 1000 cc
Time Frame: Intra-op, Post-Op
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 21 | 9
  no | 79 | 91

15. Secondary Outcome: Requirement of Cesarean Hysterectomy
Time Frame: During surgery and in the PACU (approximately 3 total hours)
Measure: Number; unit: participants
Arm/Group | Control | Uterine Cooling
Number analyzed (Participants) | 100 | 100
participants
  yes | 0 | 0
  no | 100 | 100

ADVERSE EVENTS:
Time Frame: Approximately 4 days
Description: All patients received routine post-operative and postpartum care. Their vitals were monitored for evidence of hypothermia or infection, and they received both routine post-operative day 1 labs, including a CBC, as well as follow labs as indicated. They were monitored for evidence of delayed postpartum hemorrhage.
Arm/Group | Control | Uterine Cooling
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No